CLINICAL TRIAL: NCT05642923
Title: Post-COVID-19 Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ClinAmygate (Other)
Collaborators: As-Salam Center, Maadi, Cairo, Egypt (Unknown)
Responsible Party: Principal Investigator, Emad R Issak, Dr, ClinAmygate
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR0012022
Record Dates: First submitted 2022-12-07; First posted 2022-12-08 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Post-COVID-19 Syndrome; Post-COVID Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synthetic Vitamin B1 (Active Comparator): Synthetic Vitamin B1, 400 mg per day
  Interventions: Drug: Synthetic Vitamin B1
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Synthetic Vitamin B1 — Synthetic Vitamin B1 400 mg per day
  Arms: Synthetic Vitamin B1

SUMMARY:
Fatigue is recognized as one of the most commonly presented long-term complaints in individuals previously infected with SARS-CoV-2.

DETAILED DESCRIPTION:
It has become increasingly clear that infected patients have symptoms not only in the acute phase, but also after recovery from the initial infection.

A recent meta-analysis including 4828 patients with post-COVID-19 showed that symptoms and post-acute sequelae of SARS-CoV-2 can persist weeks to months after the infection.

These patients who reported persistent symptoms have been termed "long haulers" or described as having long COVID, post-acute COVID-19, persistent COVID-19 symptoms, post COVID-19 manifestations, long-term COVID-19 effects, post-acute sequelae of COVID-19 (PASC), or post-COVID-19 syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age . 18
* Male or female
* Post-Covid-19 Fatigue

Exclusion Criteria:

* refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Fatigue scale | one month
  chalder fatigue scale: the minimum = 0 and maximum values = 33, and whether higher scores mean a worse outcome.
Fatigue scale | two month
  chalder fatigue scale: the minimum = 0 and maximum values = 33, and whether higher scores mean a worse outcome.
Fatigue scale | three month
  chalder fatigue scale: the minimum = 0 and maximum values = 33, and whether higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Incidence of adverse events | 6 months
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Asalam, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Upon request

REFERENCES:
- [Background] Jackson C. The Chalder Fatigue Scale (CFQ 11). Occup Med (Lond). 2015 Jan;65(1):86. doi: 10.1093/occmed/kqu168. No abstract available. PMID 25559796
- [Result] Kedor C, Freitag H, Meyer-Arndt L, Wittke K, Hanitsch LG, Zoller T, Steinbeis F, Haffke M, Rudolf G, Heidecker B, Bobbert T, Spranger J, Volk HD, Skurk C, Konietschke F, Paul F, Behrends U, Bellmann-Strobl J, Scheibenbogen C. A prospective observational study of post-COVID-19 chronic fatigue syndrome following the first pandemic wave in Germany and biomarkers associated with symptom severity. Nat Commun. 2022 Aug 30;13(1):5104. doi: 10.1038/s41467-022-32507-6. PMID 36042189